CLINICAL TRIAL: NCT02174159
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiretroviral Activity of MK-8507 in HIV-1 Infected Patients
Brief Title: Evaluation of Safety, Tolerability, Pharmacokinetics, and Antiretroviral Activity of Ulonivirine (MK-8507) in Human Immunodeficiency Virus (HIV-1)-Infected Participants (MK-8507-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8507-003; 2014-000660-18 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — ulonivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A: Ulonivirine 600 mg (Experimental): Single oral dose of ulonivirine 600 mg (supplied as 10 mg and 100 mg tablets) administered after an overnight fast
  Interventions: Drug: Ulonivirine
- Panel B: Ulonivirine 150 mg (Experimental): Single oral dose of ulonivirine 150 mg (supplied as 10 mg and 100 mg tablets) administered after an overnight fast
  Interventions: Drug: Ulonivirine
- Panel C: Ulonivirine <=600 mg (Experimental): Single oral dose of ulonivirine <=600 mg mg (supplied as 10 mg and 100 mg tablets) administered after an overnight fast. Inclusion of Panel C in the study, and the dose selected, will be decided pending evaluation of results for Panels A and B.
  Interventions: Drug: Ulonivirine

INTERVENTIONS:
Drug: Ulonivirine — MK-8507 administered as a single oral dose
  Other Names: MK-8507

SUMMARY:
The study will evaluate the safety, tolerability, pharmacokinetics, and antiretroviral activity of a single dose of ulonivirine in antiretroviral therapy (ART)-naive, HIV-1 infected participants. The hypothesis tested in the study is that at a safe and well-tolerated dose, ulonivirine has superior antiretroviral activity to a historical placebo control, as measured by change from baseline in plasma HIV-1 ribonucleic acid (RNA) at 168 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Male, or non-pregnant and non-breastfeeding female, or postmenopausal or surgically sterile female (confirmed with medical records, examination, or laboratory test). Male participants with female partner of childbearing potential agrees to use a medically acceptable method of contraception during the study and 90 days after receiving study drug.
* Body mass index <=35 kg/m^2
* Other than HIV infection, baseline health judged to be stable at screening and/or prior to administration of study drug
* No clinically-significant electrocardiogram abnormality
* Documented to be HIV-1 positive as determined by a positive enzyme-linked immunosorbent assay (ELISA) or quantitative polymerase chain reaction (PCR) result with confirmation
* Has a screening plasma Cluster of Differentiation (CD4) T-cell count of >200 /mm^3
* Has a plasma HIV-1 RNA >= 10,000 copies/mL within 30 days before administration of study drug
* ART-naive, defined as never having received any ART agent, or have received <=30 consecutive days of an investigational ART agent, excluding non-nucleoside reverse transcriptase inhibitors (NNRTIs), or have received <=60 consecutive days of combination ART, excluding NNRTIs
* Has not received an investigational agent or licensed ART within 30 days of study drug administration
* Diagnosed with HIV-1 infection >=3 months before screening
* Willing to receive no other ART for the duration of the study
* Has no evidence of mutations conferring resistance to NNRTIs at screening

Exclusion Criteria:

* Mentally or legally institutionalized or incapacitated, has significant emotional problems, or has a history of clinically significant psychiatric disorder
* History of clinically significant and not stably controlled abnormalities or diseases
* History of cancer, with the exceptions of 1) adequately-treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix, 2) other malignancies which have been successfully treated >=10 years before screening, or 3) participants who are highly unlikely to sustain a recurrence for the duration of the study
* History of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to drugs or food
* Positive for hepatitis B surface antigen
* History of chronic hepatitis C virus (HCV) unless there has been a documented cure or a negative HCV viral load
* Had major surgery, or donated or lost >=1 unit (~500 mL) of blood within 4 weeks before screening
* Participated in another investigational trial within 4 weeks before administration of study drug
* Unable to refrain from or anticipates the use of any medication beginning 4 weeks before administration of study drug and throughout the trial. Certain medications are permitted.
* Consumes >3 glasses of alcoholic beverages per day (1 glass is equivalent to 12 ounces of beer, 4 ounces of wine, or 1 ounce of distilled spirits). Participants who consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* Consumes >10 cigarettes per day and is unwilling to restrict smoking to <=10 cigarettes per day
* Regular user of any illicit drugs or has a history of drug abuse (including alcohol) within 2 years
* Has an immediate family member who is investigational site or sponsor staff directly involved with the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-07-16 (Actual); Study Completion 2015-07-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Plasma HIV-1 RNA | 168 hours (7 days) postdose
Number of Participants with One or More Adverse Experiences | Up to 21 days postdose

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve of Ulonivirine (AUC0-168hr) | Up to 168 hours postdose
Maximum Plasma Concentration of Ulonivirine (Cmax) | Up to 336 hours postdose
Time of Maximum Plasma Concentration of Ulonivirine (Tmax) | Up to 336 hours postdose
Plasma Concentration of Ulonivirine at 168 Hours Postdose (C168hr) | 168 hours postdose
Plasma Concentration of Ulonivirine at 336 Hours Postdose (C336hr) | 336 hours postdose
Apparent Terminal Half-Life (T1/2) of Plasma Ulonivirine | Up to 336 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Schurmann D, Jackson Rudd D, Schaeffer A, De Lepeleire I, Friedman EJ, Robberechts M, Zhang S, Liu Y, Kandala B, Keicher C, Daumer M, Hofmann J, Grobler JA, Stoch SA, Iwamoto M, Ankrom W. Single Oral Doses of MK-8507, a Novel Non-Nucleoside Reverse Transcriptase Inhibitor, Suppress HIV-1 RNA for a Week. J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):191-198. doi: 10.1097/QAI.0000000000002834. PMID 34654041